CLINICAL TRIAL: NCT06031077
Title: Effectiveness and Safety of Distal Left Transradial Access in Coronary Procedures.
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Dr. Naveen Anand Seecheran, The University of The West Indies
Other Study IDs: CREC-SA.1304/12/2021
Record Dates: First submitted 2023-07-20; First posted 2023-09-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Cardiomyopathies
Keywords: Distal Radial Artery Angiogram; Anatomical Snuff Box Angiogram
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathies | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiologist Assessed Conditions.: The consultant Cardiologist will decide on the various types of presentations and symptoms that will be use full in generating this study.
  Interventions: Procedure: cardiac catheterization

INTERVENTIONS:
Procedure: cardiac catheterization — An observational, retrospective study will be carried out. Roughly 111 patients were registered at EWMSC and Cardiac Angiograms were done via approached through the left radial access between January 2020 and June 2021 at EWMSC. However since 2021 Cardiac Angiograms were also done via the anatomical snuff box. This study seeks to compare the results of Cardiac Angiograms vs Left Radial Access and the Anatomical Snuff box.

SUMMARY:
To evaluate the effectiveness and safety of distal left radial (dLR) access in coronary procedures at a tertiary center in Trinidad and Tobago.

DETAILED DESCRIPTION:
An observational, retrospective study will be carried out. Roughly 111 patients were registered at EWMSC and Cardiac Angiograms were done via approached through the left radial access between January 2020 and June 2021 at EWMSC. However since 2021 Cardiac Angiograms were also done via the anatomical snuff box. This study seeks to compare the results of Cardiac Angiograms vs Left Radial Access and the Anatomical Snuff box.

ELIGIBILITY:
Cardiologist recommended guidelines.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caribbean decent population of Trinidad and Tobago.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of snuff box access to radial access for coronary angiography in Trinidad and Tobago. | roughly 3 years
  An observational, retrospective study will be carried out. Roughly 111 patients were registered at EWMSC and Cardiac Angiograms were done via approached through the left radial access between January 2020 and June 2021 at EWMSC. However since 2021 Cardiac Angiograms were also done via the anatomical snuff box. This study seeks to compare the results of Cardiac Angiograms vs Left Radial Access and the Anatomical Snuff box.

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Williams Medical Sciences Complex, Port of Spain, North Central, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No
The principal reason for this study is to aid physicians with the necessary data to perform cardiac catherisation and to show them different access points.